CLINICAL TRIAL: NCT06245538
Title: Acute Effects of Physical Exercise of Different Intensities on Biological and Psychological Outcomes Under Subclinical Stress and in Health
Brief Title: Exercise Intensity on Brain & Mental Health in Stress
Acronym: ExStress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: The Knowledge Foundation (Unknown); Avonova (Unknown); SATS (Unknown); Itrim (Unknown)
Responsible Party: Principal Investigator, Maria Ekblom, Professor, The Swedish School of Sport and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2022-07297-01; 2023-08181-02 (Other: Swedish ethical review authority)
Record Dates: First submitted 2024-01-28; First posted 2024-02-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults; Adults With Stress-related Symptoms
Keywords: FNIRS; Neuroplasticity; Neuroinflammation; cerebral blood flow; Exercise intensity; Psychological stress
MeSH Terms: conditions — Neuroinflammatory Diseases; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized-order crossover experimental trial with three experimental conditions separated by a wash-out period of 7 days: 20-min leg cycling exercise at moderate intensity, 20-min leg cycling exercise at vigorous intensity, and 20-min seated rest (passive control condition)
Masking Description: The outcomes assessors follow standard operation procedures with automatic analyses and are blinded to study condition and individual stress ratings when analysing the collected data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seated rest (Experimental): Participants will be resting while seated on a comfortable chair for 20 minutes
  Interventions: Behavioral: Seated rest
- Exercise at moderate intensity (Experimental): Participants will perform a 20-min leg cycling exercise on a cycle ergometer at moderate intensity (60% of VO2max)
  Interventions: Behavioral: Exercise at moderate intensity
- Exercise at vigorous intensity (Experimental): Participants will perform a 20-min leg cycling exercise on a cycle ergometer at vigorous intensity (80% of VO2max)
  Interventions: Behavioral: Exercise at vigorous intensity

INTERVENTIONS:
Behavioral: Seated rest — Participants will be resting while seated on a comfortable chair for 20 minutes
  Arms: Seated rest
Behavioral: Exercise at moderate intensity — Participants will perform a 20-min leg cycling exercise on a cycle ergometer at moderate intensity (60% of VO2max)
  Arms: Exercise at moderate intensity
Behavioral: Exercise at vigorous intensity — Participants will perform a 20-min leg cycling exercise on a cycle ergometer at vigorous intensity (80% of VO2max)
  Arms: Exercise at vigorous intensity

SUMMARY:
This study aims to examine the role of exercise intensity in the acute effects of a single bout of aerobic exercise on neurotrophic factors, biomarkers of stress and inflammation, working memory task-related changes in prefrontal cortex oxygenation in adults with sub-clinical levels of stress-related symptoms.

DETAILED DESCRIPTION:
This study initially set out to include 43 adult (20 - 40 years) participants experiencing stress-related symptoms and 43 healthy controls, matched by age, sex, and fitness. These procedures were approved by the Swedish Ethical Review Autority (Approval number 2022-07297-01 and 2023-08181-02). Due to recruitment difficulties the design was later changed to include all individuals with sub-clinical stress symptoms and using stress as a covariate instead of comparing groups of healthy and stressed individuals (Ethical review approval number 2025-01786-02). This is a randomized-order crossover experimental trial with three experimental conditions separated by a wash-out period of 7 days: 20-min leg cycling exercise at moderate intensity, 20-min leg cycling exercise at vigorous intensity, and 20-min seated rest (passive control condition).

Prior to entering the study, study inclusion/exclusion criteria will be controlled using digital screening. Before the experimental sessions, all participants will complete two introductory study visits. At the first introductory visit, the participant's maximal oxygen uptake (VO2max) will be determined using a fitness test. This information will be used to determine the individual workloads (% of individual VO2max) that the participant will be cycling at during the experimental session. At the second introductory visit, participants will complete a familiarization session, in which key methodological aspects of the study will be introduced to participants. Participants' augmentation index, as a measure of arterial stiffness, will also be completed during this visit.

In each of the three experimental sessions, participants will perform a computerized working memory task (n-back task) pre- and post-exercise (or seated rest). During the working memory task, functional near-infrared spectroscopy (fNIRS) will be used to measure task-related changes in prefrontal cortex oxygenation. As such, each participant will complete six fNIRS measurements, two measurements (pre, post) for each of the three experimental sessions (moderate, high, control). Simultaneous with the fNIRS measurements, blood flow velocity in the left and right middle cerebral artery will be assessed during the n-back tasks using Transcranial Doppler ultrasound. At each experimental session, blood will also be sampled from the antecubital vein at six time points: pre the first n-back task, pre and post the cycling exercise (or seated rest), pre and post the second n-back task, and post the final 10-min seated rest. Whole blood samples will be assessed for blood gases, acid-base status, electrolytes, hematocrit level, platelet count, and glucose. The separated blood plasma and serum samples will be used for measurements of neurotrophic factors, lactate, biomarkers of stress and inflammation, and factors involved in blood glucose control. Blood samples will also be used for targeted DNA screening for alleles of the BDNF.

Additionally, the participant's current mood, mental and physical fatigue, heart rate variability (HRV) and blood pressure will be assessed during four 10-min seated rest periods: pre and post n-back, and pre and post cycling exercise (or seated rest). Prior to each experimental study session, participants will have assessments of sleep quality the night before, current health status, physical activity level during the week prior to the test day, sleepiness level the last 10 min, and current mood. Participant's sleep quality and heart rate variability during the night before and after each experimental session will also be assessed.

A release of an updated version of this study was attempted prior to completion of the study on October 3 2025, but due to a shutdown of the US goverment this was not possible to register until in November 24 2025.

ELIGIBILITY:
Inclusion Criteria:

Participants experiencing sub-clinical levels of stress-related symptoms:

* Age: 20-40 years
* Absence of contraindications to physical exercise
* Do not participate in any other study
* Total score on the self-assessment scale 4-factor Shirom-Melamed Burnout Measure-19 lower than or equal to 4.00

Exclusion Criteria:

* Medical contraindication to catheterization of the antecubital vein and blood sampling
* Dementia
* Alcohol abuse
* Smoking
* Chronic medication that is considered to affect study outcomes
* Chronic disease/syndrome such as migraine, fibromyalgia, chronic fatigue syndrome, bipolar syndrome, high blood pressure, cardiovascular disease, chronic obstructive pulmonary disease (COPD) or other lung disease
* Post-COVID
* Other somatic diseases, disorders, or injuries that may affect the physical ability during physical exercise

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral blood flow in prefrontal cortex | from before to after 20 minutes of exercise or seated rest
  working memory task-related changes in prefrontal cortex oxygenation measured using functional near-infrared spectroscopy

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  pro and mature BDNF in blood sample taken from the forearm antecubital vein; concentrations measured in blood plasma and serum
Working memory performance | At one time point before and one time point after 20 minutes of exercise or seated rest (In total over 1 hour)
  computerized working memory task (n-back: 1-, 2- and 3-back)
DNA allele of brain-derived neurotrophic factor | At one time point at baseline
  in blood sample taken before intervention from the forearm antecubital vein
Platelet count | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  in blood sample taken from the forearm antecubital vein
Cortisol | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  biomarker of stress; in blood sample taken from the forearm antecubital vein
Epinephrine | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  biomarker of stress; in blood sample taken from the forearm antecubital vein
Norepinephrine | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  biomarker of stress; in blood sample taken from the forearm antecubital vein
C-reactive protein (CRP) | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  as a measure of systemic inflammation; in blood sample taken from the forearm antecubital vein
Interleukin 6 (IL-6) | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  as a measure of systemic inflammation; in blood sample taken from the forearm antecubital vein
Tumor necrosis factor alpha (TNF-α) | At three time points before and four time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  as a measure of systemic inflammation; in blood sample taken from the forearm antecubital vein
Mood | At two time points before and two time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  measured with a short version of Positive and Negative Affect Schedule (PANAS-SF) that include 5 positive and 5 negative affect states; the scoring scale is from 1 (very slightly or not at all) to 5 (extremely)
Mental fatigue | At two time points before and two time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  measured using Visual Analogue Scale (VAS-F); scoring scale: a line with 100 mm in length with scores falling between 0 mm (extremely alert) and 100 mm (extremely tired)
Physical fatigue | At two time points before and two time points after 20 minutes of exercise or seated rest (In total over 2 hours)
  measured using Borg Rating of Perceived Exertion scale; scoring scale: from 6 (no exertion) to 20 (maximal exertion)
Sleep quality | Over the night before and the night after each experimental session (In total over 36 hours)
  measured using a Single-Item Sleep Quality Scale; scoring scale is from 0 (terrible) to 10 (excellent)
Sleepiness | At single time point before 20 minutes of exercise or seated rest
  measured using Karolinska Sleepiness Scale; scoring scale is from 1 (extremely alert) to 9 (extremely sleepy)
Heart rate variability | Over the night before and the night after each experimental session (In total over 36 hours)
  as an additional indicator of stress-related symptoms; measured with heart rate sensor and monitor
Augmentation index | At a single time point at baseline
  as a measure of arterial stiffness and indicator of cardiovascular health

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ekblom, PhD, Principal Investigator — The Swedish School of Sport and Health Sciences (GIH)
Locations (1):
- The Swedish School of Sport and Health Sciences, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make individual participant data available to other researchers.